CLINICAL TRIAL: NCT07087678
Title: A Prospective, Randomised, Open Label Feasibility Trial Comparing BurstDR Microdosing Versus Tonic Occipital Nerve Stimulation for Patients With Refractory Chronic Migraine
Brief Title: Occipital Nerve Stimulation in Chronic Migraine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 321114
Record Dates: First submitted 2025-04-30; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Chronic Migraine, Headache; Refractory Migraine
Keywords: Chronic migraine; Occipital nerve stimulation; BurstDR microdosing; Refractory migraine
MeSH Terms: conditions — Headache; Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Eligible subjects will complete a baseline headache diary and questionnaires, and then be randomised to BurstDR microdosing or tonic stimulation. After implantation and stabilisation, the device is activated and they continue to complete headache diary and questionnaires at 1 month, 3 months and 6 months whilst further programming optimisation occurs. Non-responders are offered the opportunity to cross over into the opposite arm. Further diary and questionnaire monitoring will occur at 1 year and optional long term follow up at 2 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ONS using tonic stimulation with Prodigy Internal Pulse Generator (Active Comparator): Tonic stimulation provides continuous electrical stimulation with perceptible paraesthesia to the occipital region. It is the standard of care at present in this unit and in most published studies of ONS.
  Interventions: Device: Prodigy internal pulse generator occipital nerve stimulator
- ONS using BurstDR microdosing stimulation with Prodigy Internal Pulse Generator (Experimental): BurstDR microdosing provides pulses of stimulation at a lower amplitude but higher frequency and a larger pulse width than Tonic stimulation. The stimulation is not perceptible to the patient and there is no paraesthesia. Early reports of spinal cord stimulation and suggest it may be preferable for patients and does not have any serious adverse effects.
  Interventions: Device: Prodigy internal pulse generator occipital nerve stimulator

INTERVENTIONS:
Device: Prodigy internal pulse generator occipital nerve stimulator — Electrical stimulation of the occipital nerves using an implantable device

SUMMARY:
The goal of this clinical trial is to compare two different types of occipital nerve stimulation (BurstDR (dorsal root) microdosing versus Tonic) in chronic refractory migraine. The main questions it aims to answer is whether BurstDR microdosing is effective in reducing moderate to severe headache days compared to Tonic stimulation (which is currently in use). Additionally, the safety of both types of stimulation will be studied.

Participants will be asked to keep a headache diary, then have the device implanted and programmed, and keep a subsequent headache diary to see if there is an improvement in their headaches after three moths of stimulation. If they don't respond to treatment, they will be allowed to swap to the other type of stimulation to see if this improves their symptoms.

DETAILED DESCRIPTION:
Eligible subjects will complete a baseline headache diary and questionnaires, and then be randomised to BurstDR microdosing or tonic stimulation. After implantation and stabilisation, the device is activated and they continue to complete headache diary and questionnaires at 1 month, 3 months and 6 months whilst further programming optimisation occurs. Non-responders are offered the opportunity to cross over into the opposite arm. Further diary and questionnaire monitoring will occur at 1 year and optional long term follow up at 2 years.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years old and diagnosed with intractable chronic migraine by a headache specialist, as defined by the International Classification of Headache Disorders-3 (ICHD-3).

Subject should have failed to gain benefit from at least 4 classes of oral preventative medications, Botulinum toxin or acupuncture as defined by NHS (National Health Service) England Subject has been diagnosed at least 6 months prior to study enrolment with migraine headache with or without aura according to the ICHD-3 criteria 1.1, 1.2.1, or 1.3.

Subject is able to distinguish migraine attacks from other headaches (e.g. tension type headache, cluster headaches).

Subject agrees to not participate in supplemental or alternative therapy through the Follow Up Period of the study. This includes acupuncture, spinal manipulation, TENS (transcutaneous electrical nerve stimulation), and magnetic fields treatments.

Subject has the ability to read, comprehend, and to reliably record information as required by the Protocol.

Subject is able to provide written informed consent prior to participation in the study.

Exclusion Criteria:

Subject's overall health, age and/or comorbidities place subject at high risk for complications from surgery and/or general anaesthesia.

Subject has clinically significant drug (including opioid) or alcohol abuse as defined by DSM-IV-TR (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision), will likely be unable to refrain from substance abuse throughout the study, has another significant pain problem, substance abuse or active depressive episode that might confound the study assessments in the opinion of the Investigator.

Subject is currently participating or has participated in the last month in another clinical study in which the subject has, is, or will be exposed to, an investigational drug or device, except for sponsor-related studies.

Subject is felt to be at risk of non-compliance (e.g., for completing the diary/questionnaires or returning for required follow-up visits) in the Investigator's opinion.

Subject has medication overuse headache which has not been managed (by withdrawal of the causative medication).

Subject is a woman of childbearing potential who is pregnant, nursing, or not using effective contraception.

Subject has an active implantable device such as pacemaker/ defibrillator or other neurostimulation device.

Subject has a history of bleeding disorders or coagulopathy or is unable to discontinue anticoagulation, antiplatelet, or GP (glycoprotein) IIb IIIa inhibitor medication in preparation for the implantation procedure.

Subject is not suitable for the study for any reason in the judgment of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of ONS | 3 months post activation of ONS
  The primary objective is to compare the reduction in moderate to severe headache days at three months (i.e. weeks 8-12 post activation of the ONS device) in patients who have tonic stimulation compared to those having BurstDR stimulation.
  Severity of headache will be recorded on a 0-10 pain scale in a daily in a headache diary which is completed by the patient throughout the baseline and intervention period.
  Moderate to severe headache days are defined as: a 24-hour period with headache pain of moderate or severe intensity that lasts at least 4 hours without medication, or a day with a headache pain of at least moderate intensity that responds to acute treatment with a migraine-specific medication. On the pain scale, 1-3/10 equates to mild pain, 4-6/10 equates to moderate pain and 7-10/10 equates to severe pain.

SECONDARY OUTCOMES:
Number and severity of adverse events with Tonic and BurstDR stimulation | 1,3,6 months compared to baseline
  Adverse events (AEs) will be recorded for all patients at each follow up appointment (and in between appointments if appropriate).
  Each adverse event will be assessed for severity, causality, seriousness and expectedness. AEs will be recored from the time of ONS insertion until the end of the subject's involvement in the trial.
  Definitions:
  Mild AE: does not interfere with the participant's daily routine, and does not require further intervention; it causes slight discomfort
  Moderate AE: interferes with some aspects of the participant's routine, or requires further intervention, but is not damaging to health; it causes moderate discomfort
  Severe AE: results in alteration, discomfort or disability which is clearly damaging to health
30% responder rate | 1,3,6 months compared to baseline
  The proportion of subjects which achieve ≥30% reduction in headache load at one, three and six months compared to baseline) for tonic verses BurstDR microdosing
Monthly migraine days | 1,3,6 months compared to baseline
  Change in monthly migraine days
Monthly moderate to severe headache days | 6,9,12 months post activation
  Change in monthly moderate to severe headache days compared to baseline
Headache severity | 1,3,6 months compared to baseline
  Change in monthly mean headache severity compared to baseline
  The pain scale described in the primary outcome measure will be applied here.
Change in mean monthly headache load | At 1, 3, 6 months post activation
  Headache load is calculated as the sum of the product of pain severity (on 0-10 scale), headache duration in hours for each attack over a 28 day period.
  A lower headache load equates to a better outcome.
HIT-6 score (Headache Impact Test - 6) | 1,3 and 6 months post activation
  Change in mean HIT-6 score compared to baseline
  A lower HIT-6 score equates to a better outcome. The minimum value is 36 and the maximum value is 78.
MIDAS (migraine disability assessment) score | 1,3 and 6 months post activation
  Change in MIDAS score compared to baseline
  A lower score equates to a better outcome. The minimum value is 0 and the maximum value is 270.
Hospital anxiety scores (HADS-A) | 1,3 and 6 months post activation
  Change in HADS-A compared to baseline A lower score equates to a better outcome. The minimum score is 0 and the maximum is 21.
Hospital depression score (HADS-D) | 1,3 and 6 months post activation
  Change in HADS-D compared to baseline
  A lower score equates to a better outcome. The minimum score is 0 and the maximum is 21.
Change in EuroQol-5D5L (European Quality of Life 5 Dimensions) score | 1,3,6 months compared to baseline
  The EuroQol-5D5DL score measures quality of life in dimensions of life activities, and includes a global rating of their overall health.

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant-level dataset may be made available on request for clinical or academic purposes only, after publication of the trial results.